CLINICAL TRIAL: NCT06124885
Title: Real-time Early Detection of Nephrotoxicity by Accurate and Faster Urinary Biomarker Analysis With SeroFlow Technology (RenaFAST Study)
Brief Title: Real-time Early Detection of Nephrotoxicity by Urinary Biomarker Analysis With SeroFlow Technology
Acronym: RenaFAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021/00920
Record Dates: First submitted 2023-10-16; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-06

CONDITIONS: Acute Kidney Injury
Keywords: Nephrotoxicity; Urinary biomarkers; Clusterin; monocyte chemoattractant protein-1 (MCP1); Beta-2 microglobulin (ß2MG); Anti-microbials; Calcineurin inhibitors
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Single arm design. All eligible and consenting patients will have their time-point urine samples collected and biomarker levels measured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AKI risk screening using RenaFAST POCT test kits (Experimental): All consenting patients will have a real-time biomarker analysis done at 5 time-points during their course of drug therapy using the renaFAST kits.
  Interventions: Diagnostic Test: AKI risk screening using RenaFAST POCT test kits

INTERVENTIONS:
Diagnostic Test: AKI risk screening using RenaFAST POCT test kits — Based on the type and duration of drug therapy, a maximum of 5 time-point urine samples will be collected and real-time biomarker measurement will be done using the RenaFAST POCT kits. Additionally, Trefoil factor 3 (TFF3) biomarker levels will also be quantified using developed POCT kits.
  Patients with all 3 biomarker (Clusterin, MCP1 and ß2MG) levels higher than the study cut-off will be identified as high-risk for AKI. The nephrology consultants within the research team will perform a medical chart and physical review (where required) of these patients, detailing potential actions to be taken in research data collection forms. No actual intervention (other than a patient review) will be performed.

SUMMARY:
The study aims to perform real-time validation of the RenaFAST kit (a point-of-care test kit that quantifies three urinary proteins) in predicting acute kidney injury(AKI) among patients prescribed drug therapies of nephrotoxic potential. Based on the type and duration of drug therapy, a maximum of 5 time-point urine samples will be collected from consenting patients and a real-time biomarker analysis will be conducted using the RenaFAST kits.

DETAILED DESCRIPTION:
All eligible patients who fulfill the inclusion and exclusion criteria will be approached for consent. The patients with the highest AKI risk (with all 3 urine biomarkers, Clusterin, monocyte chemoattractant protein-1 (MCP1), and Beta-2 microglobulin (ß2MG), above prediction threshold set by the study) will be identified. The nephrology consultants within the research team will perform a medical chart and physical review(where required) of these patients, noting potential actions to be taken in data collection forms. This will help in evaluating if indeed there are perceived interventions that could potentially be delivered in response to early prediction of AKI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive a projected ≥7 days of therapy of antimicrobials including aminoglycosides (i.e., gentamicin or amikacin), vancomycin, polymyxin, amphotericin and foscarnet.
* Patients who receive a projected ≥7 days of Calcineurin inhibitors (cyclosporin, tacrolimus)
* Patients who receive a projected ≥7 days of anti-virals (Cidofovir and Ganciclovir)
* Patients who receive Anti-cancer drugs (Chemotherapy such as cisplatin, Ifosfamide, Methotrexate, Pemetrexed) or
* Patients who receive Anti-cancer drugs (Immunotherapy such as immune checkpoint inhibitors as well as types of VGEF inhibitors that are associated with acute kidney injury)

Exclusion Criteria:

* Patients with AKI prior to therapy initiation.
* Patients with baseline eGFR < 15 mL/min/1.73m2 (stage 5 chronic kidney disease)
* Patients admitted to intensive care unit at study baseline, as critical illness is a natural confounder to AKI
* Females who are pregnant
* Immediate post-kidney transplant recipients (initial 3 months following transplant).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Presence of an Acute kidney injury (AKI) event | Start date of drug therapy till one week post end date of drug therapy
  AKI will be defined by the minimum stage 1 criterion in accordance to KDIGO AKI criteria:
  1. Relative increase in serum creatinine of 1.5 times or higher, versus the baseline.
  2. Absolute increase in serum creatinine of > 26.5 μmol/L within 48 hours.
  Additionally, for those administered cisplatin, cases of severe hyponatremia needing hospitalization for severe dehydration and intravenous fluid-rescue will also be taken as an outcome measure of clinically-evident kidney injury and renal salt wasting.
  If the subject meets any one of the above 3 criteria, the patient will be recorded as having suffered an AKI event.

SECONDARY OUTCOMES:
Severity of AKI event | From the date of AKI onset to date of peak AKI
  Peak AKI severity will be determined by highest recorded serum creatinine levels of patient.
Number of AKI days till recovery | From the date of AKI onset to date of resolution of AKI
  Number of days from the onset of AKI (as per aforementioned AKI criteria) to resolution of AKI (Defined as when serum creatinine levels reach baseline levels or no longer meet the AKI criterion, whichever is earlier)
Length of stay in hospital | From the date of admission to the date of discharge of patient from hospital, assessed up to 12months from date of consent
  Duration of hospital stay will be determined based on admission and discharge dates of the patient, for the period relevant to study participation.
Number of patients requiring dialysis treatment for the AKI event | From the date of AKI onset to date of resolution of AKI
  Whether patient required dialysis/CRRT for treatment of AKI event

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Ruey Dr Chua, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Da Y, Akalya K, Murali T, Vathsala A, Tan CS, Low S, Lim HN, Teo BW, Lau T, Ong L, Chua HR. Serial Quantification of Urinary Protein Biomarkers to Predict Drug-induced Acute Kidney Injury. Curr Drug Metab. 2019;20(8):656-664. doi: 10.2174/1389200220666190711114504. PMID 31296157